CLINICAL TRIAL: NCT05431101
Title: Absorbable Versus Non-absorbable Sutures for Wound Closure in Carpal Tunnel Release: a Randomized Controlled Trial
Brief Title: abSorbable vErsus Non-absorbable SuturEs for Wound Closure in Carpal Tunnel Release
Acronym: SENSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gelre Hospitals (Other)
Collaborators: Deventer Ziekenhuis (Other)
Responsible Party: Principal Investigator, Pauline Verhaegen, Doctor, Gelre Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/551
Record Dates: First submitted 2022-06-21; First posted 2022-06-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Carpal Tunnel Syndrome; Wound Infection; Suture, Complication
Keywords: carpal tunnel syndrome; wound infection; absorbable sutures; non-absorbable sutures
MeSH Terms: conditions — Carpal Tunnel Syndrome; Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Absorbable sutures (Active Comparator): Absorbable sutures Vicryl rapide or Safil quick
  Interventions: Procedure: Carpal Tunnel Release
- Non-absorbable sutures (Active Comparator): Non-absorbable sutures Ethilon or Flexocrin
  Interventions: Procedure: Carpal Tunnel Release

INTERVENTIONS:
Procedure: Carpal Tunnel Release — Transection of flexor retinaculum for patients who have carpal tunnel syndrome

SUMMARY:
Carpal Tunnel Syndrome is a prevalent condition, up to 9% in women and 0.6% in men. Surgical decompression in the most effective treatment. After surgery, approximately 1,8% of the patients develop a wound infection. Possibly, the type of sutures used can influence the prevalence of wound infection. In this RCT the incidence of infection is investigated between the use of absorbable versus non-absorbable sutures in carpal tunnel release.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome is a prevalent condition; up to 9% in women and 0.6% in men. It causes complaints of paresthesia, pain, numbness and loss of strength. Surgical decompression is the most effective treatment. After surgery, approximately 1,8% of the patients develop a wound infection. Possibly, the type of suture material which is used can influence the prevalence of wound infection. In current clinical practice both absorbable and non absorbable sutures are used. In literature, various hypothesis are described: Absorbable sutures could give more reaction of macrophages and therefore a higher chance on infection. This would not be the case for non-absorbable sutures, since they will be removed. However, in literature, there is still not enough evidence for superiority of absorbable or non-absorbable suture. In this RCT the incidence of infection is investigated between the use of absorbable versus non-absorbable sutures in carpal tunnel release.

The primary outcome is the ASEPSIS wound score. This will be scored by independent investigators.

Use of antibiotics, handtherapy and extra outpatient visits will be recorded.

Patients are asked to register their NRS scores the first three weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

• indication for carpal tunnel release

Exclusion Criteria:

* carpal tunnel syndrome which has yet been operated
* injection with corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2604 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
ASEPSIS wound score (Additional treatment, Serous discharge, Erythema, Purulent exudate, Separation of deep tissues, Isolation of bacteria, and Stay as inpatient prolonged over 14 days) | 10 to 14 days post surgery
  score based on a picture made of the wound 10-14 days post carpal tunnel release. Minimum score 0, maximum score 70, score above 40 is categorized as wound infection

SECONDARY OUTCOMES:
NRS score (Numeric Rating Scale for pain) | until three weeks post surgery
  pain score, minimum score 0, maximum score 10. Unbearable pain is scored as 10, no pain is scored as 0.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Gelre Ziekenhuizen, Apeldoorn
  - Deventer Ziekenhuis, Deventer